CLINICAL TRIAL: NCT03222245
Title: The Effect of Injectable Therapies on Health Status, Quality of Life and Treatment Satisfaction in Patients With Type 2 Diabetes: Prospective Observational Cohort Study
Brief Title: The Effect of Injectable Therapies on Quality of Life in Diabetes
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: V5.0
Record Dates: First submitted 2017-07-14; First posted 2017-07-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: This group consists of participants identified as needing to start injectable therapy within 1 month from the recruitment date (50% insulin and 50% GLP-1 analogues)
- Non-exposed group: This group consists of participants treated with oral anti- hyperglycaemic agents (OAHAs) and their combinations

SUMMARY:
This study is only open to sites in the Wessex CRN. The aim of diabetes treatment is to achieve and maintain as optimal blood glucose levels as possible to prevent unpleasant symptoms associated with high blood sugars and long-term complications of diabetes. This can be achieved with oral tablets, subcutaneous injectable diabetes therapies such as insulin or GLP-1 analogues.

Injectable therapies can significantly improve glucose control, but the counter to this might be an increased treatment burden, patient and clinician's inertia to initiate injectable treatments and the potential side effects of the medications.

These treatment aspects may critically affect patients' health related quality of life and satisfaction with treatment which can powerfully influence patients' compliance and self-management behaviours. This is an observational cohort study and its overall aim is to compare the health status, quality of life (QOL) and treatment satisfaction in two cohorts of patients with type 2 diabetes - those treated with oral diabetes drugs (nonexposed group) and those on subcutaneous injectable therapies (exposed group).

The changes in the above parameters will be measured by applying three questionnaires to both groups of participants at baseline and after 6 months of treatment:

1. ADDQoL measures diabetes specific quality of life
2. DTSQ measures treatment satisfaction
3. SF-36 measures overall health status

Study duration is six months for each participant and over this period participants will receive three telephone or face to face contacts (based on their preference) with the research team. The questionnaires will be posted to participants at baseline and at 6 months and will be completed in paper form and returned to research team in pre-paid selfaddressed envelopes.

It is hoped that this study will provide valuable understanding of the effect of injectable therapies on QOL and treatment satisfaction in our local population with type 2 diabetes which can then be carefully factored into clinical decisions when initiating or intensifying diabetes treatments.

DETAILED DESCRIPTION:
The aim of diabetes treatment is to achieve and maintain as optimal blood glucose levels as possible to prevent unpleasant symptoms associated with high blood sugars and long-term complications of diabetes. This can be achieved with oral tablets, subcutaneous injectable diabetes therapies such as insulin or GLP-1 analogues.

Injectable therapies can significantly improve glucose control, but the counter to this might be an increased treatment burden, patient and clinician's inertia to initiate injectable treatments and the potential side effects of the medications.

These treatment aspects may critically affect patients' health related quality of life and satisfaction with treatment which can powerfully influence patients' compliance and self-management behaviours. This is an observational cohort study and its overall aim is to compare the health status, quality of life (QOL) and treatment satisfaction in two cohorts of patients with type 2 diabetes - those treated with oral diabetes drugs (nonexposed group) and those on subcutaneous injectable therapies (exposed group).

The changes in the above parameters will be measured by applying three questionnaires to both groups of participants at baseline and after 6 months of treatment:

1. ADDQoL measures diabetes specific quality of life
2. DTSQ measures treatment satisfaction
3. SF-36 measures overall health status

Study duration is six months for each participant and over this period participants will receive three telephone or face to face contacts (based on their preference) with the research team. The questionnaires will be posted to participants at baseline and at 6 months and will be completed in paper form and returned to research team in pre-paid selfaddressed envelopes.

It is hoped that this study will provide valuable understanding of the effect of injectable therapies on QOL and treatment satisfaction in our local population with type 2 diabetes which can then be carefully factored into clinical decisions when initiating or intensifying diabetes treatments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a coded diagnosis of type 2 diabetes diagnosed at least 1 year prior to start of the study to minimise bias present from psychological effect of diagnosis
* Age 18 y inclusive and above
* Participant is willing and able to give informed consent for participation in the study
* Participants currently treated with OAHAs and their combinations
* Completely naïve to self-administration of sc injections as part of diabetes treatment or for any other medical condition
* Exposed group will consist of participants identified as needing to start and starting sc injectable therapy (insulin or GPL-1 analogue) within 1 month of recruitment.
* Non-exposed group will consist of participants managed with diet or OAHA therapies and their combinations, who require an addition of a new OAHA to their current therapy to intensify their diabetes control

Exclusion Criteria:

* Current diagnosis means that their predicted lifespan is shorter than duration of the study
* Medical condition that may affect participants' quality of life eg diagnosis of cancer, undergoing chemotherapy
* History of or current diagnosis of depression
* Planning of moving out of area before completion of the study
* Pregnant and intention of becoming pregnant
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local population of patients with type 2 diabetes from both the primary and secondary care setting.
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | 26 weeks
  Change in ADDQoL score Change in DTSQ score

SECONDARY OUTCOMES:
Change in HbA1c | 26 weeks
  Change in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allard, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospital NHS Trust, Portsmouth, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No